CLINICAL TRIAL: NCT01054404
Title: The Effect of Furosemide Versus Placebo on Brain Relaxation and Incidence of Significant Intravascular Volume Depletion in Human Subjects Receiving Mannitol
Brief Title: Furosemide vs Placebo for Brain Relaxation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Concern for volume depletion and electrolyte abnormalities in furosemide arm.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Bebawy, Assistant Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00016126
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Brain Swelling; Brain Edema; Dehydration
Keywords: Brain Swelling; Brain Edema; Dehydration
MeSH Terms: conditions — Brain Edema; Dehydration | interventions — Furosemide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide (Active Comparator): Furosemide 0.3 mg/kg
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator): Up to 5 mL saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Furosemide — Furosemide 0.3 mg/kg
  Other Names: Lasix
  Arms: Furosemide
Drug: Placebo — Placebo (up to 5mL)
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Increased brain bulk may be problematic during brain surgery for tumors because it may limit surgical exposure and access to the surgical site. Mannitol, an osmotic diuretic, is commonly given to alleviate brain bulk, and sometimes furosemide in a small dose is added if mannitol alone is insufficient. It is unclear if adding this furosemide truly helps to diminish brain bulk, and it is possible that furosemide may cause too much diuresis, leading to dehydration and its side effects (e.g., low blood pressure). Our purpose is to investigate what the effects of furosemide are in the setting of brain surgery for tumors, specifically with regards to decreasing brain bulk and/or causing dehydration.

Study Hypothesis: The addition of furosemide to mannitol will result in improved brain relaxation in human subjects undergoing craniotomy for brain tumor resection than that seen with mannitol alone. However, the combination of mannitol and furosemide will also lead to more significant intravascular volume depletion than that seen with mannitol alone.

DETAILED DESCRIPTION:
Rating of brain relaxation will be on a 4-point scale:

0 = brain very relaxed under dura, acceptable

1. = brain adequately relaxed under dura, acceptable
2. = brain slightly tense under dura, acceptable
3. = brain very tense under bulging dura, unacceptable

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include:

  * ASA PS I-III
  * Age 18 or older
  * Presenting for elective resection of primary or metastatic supratentorial brain tumor(s)

Exclusion Criteria:

* • ASA PS IV or V

  * Age less than 18
  * Emergency surgery due to severely elevated ICP/impending brainstem herniation
  * Concurrent use of diuretics for any indication
  * Infratentorial/posterior fossa/cerebellar tumor resection
  * Moderate/severe cardiac disease with limitation in contractility as measured by preoperative echocardiogram (EF < 30%)
  * Severe pulmonary hypertension as measured and/or observed by preoperative studies
  * Preoperative use of steroids (within 6 months, including those on standing doses)
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Bebawy, MD, Principal Investigator — Northwestern University; Dhanesh K Gupta, MD, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Thenuwara K, Todd MM, Brian JE Jr. Effect of mannitol and furosemide on plasma osmolality and brain water. Anesthesiology. 2002 Feb;96(2):416-21. doi: 10.1097/00000542-200202000-00029. PMID 11818776
- [Background] Todd MM, Cutkomp J, Brian JE. Influence of mannitol and furosemide, alone and in combination, on brain water content after fluid percussion injury. Anesthesiology. 2006 Dec;105(6):1176-81. doi: 10.1097/00000542-200612000-00017. PMID 17122580
- [Background] Rudehill A, Lagerkranser M, Lindquist C, Gordon E. Effects of mannitol on blood volume and central hemodynamics in patients undergoing cerebral aneurysm surgery. Anesth Analg. 1983 Oct;62(10):875-80. PMID 6412595
- [Background] Todd MM, Warner DS, Sokoll MD, Maktabi MA, Hindman BJ, Scamman FL, Kirschner J. A prospective, comparative trial of three anesthetics for elective supratentorial craniotomy. Propofol/fentanyl, isoflurane/nitrous oxide, and fentanyl/nitrous oxide. Anesthesiology. 1993 Jun;78(6):1005-20. doi: 10.1097/00000542-199306000-00002. PMID 8512094
- [Background] Rozet I, Tontisirin N, Muangman S, Vavilala MS, Souter MJ, Lee LA, Kincaid MS, Britz GW, Lam AM. Effect of equiosmolar solutions of mannitol versus hypertonic saline on intraoperative brain relaxation and electrolyte balance. Anesthesiology. 2007 Nov;107(5):697-704. doi: 10.1097/01.anes.0000286980.92759.94. PMID 18073543

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 patients enrolled sequentially, no dropouts
Groups:
- Furosemide: Furosemide : Furosemide 0.3 mg/kg
- Placebo: Placebo : Placebo (up to 5mL)
Period: Overall Study
Arm/Group | Furosemide | Placebo
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide | Placebo | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 2 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (16.6) | 52.1 (15.6) | 51.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Acceptable vs. Unacceptable Brain Relaxation at Dural Opening
Description: Rating of brain relaxation will be on a 4-point scale:
  0 = brain very relaxed under dura, acceptable
  1. = brain adequately relaxed under dura, acceptable
  2. = brain slightly tense under dura, acceptable
  3. = brain very tense under bulging dura, unacceptable
Time Frame: just prior to dural opening for each subject
Measure: Mean (Standard Error); unit: units on a scale 0-3
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 10 | 13
units on a scale 0-3 | 1.5 (.17) | 1.3 (.13)

ADVERSE EVENTS:
Arm/Group | Furosemide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13

LIMITATIONS AND CAVEATS:
Recruitment was stopped at 23 subjects because of concern that the administration of furosemide was producing such a large diuresis that clinically significant and potentially unsafe hypovolemia and electrolyte abnormalities were developing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No